CLINICAL TRIAL: NCT03074656
Title: A NORwegian Multicentre Randomised Controlled Trial Assessing the Effectiveness of Tailoring Infliximab Treatment by Therapeutic DRUg Monitoring - The NOR-DRUM Study
Brief Title: The Norwegian Drug Monitoring Study
Acronym: NOR-DRUM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diakonhjemmet Hospital (Other)
Collaborators: Oslo University Hospital (Other); University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Espen A. Haavardsholm, MD PhD, Professor, MD, PhD, Diakonhjemmet Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DIA2016-1
Record Dates: First submitted 2017-02-10; First posted 2017-03-09 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Rheumatoid Arthritis; Spondyloarthritis; Ankylosing Spondylitis; Crohn Disease; Ulcerative Colitis; Psoriasis; Psoriatic Arthritis
Keywords: infliximab; therapeutic drug monitoring; anti drug antibodies; TDM
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylarthritis; Spondylitis, Ankylosing; Crohn Disease; Colitis, Ulcerative; Psoriasis; Arthritis, Psoriatic | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Therapeutic drug monitoring (Experimental): Administration of infliximab according to a treatment strategy based on therapeutic drug monitoring and assessments of anti-drug antibodies
  Interventions: Other: Therapeutic drug monitoring
- Standard care (Active Comparator): Administration of infliximab according to standard clinical care, without knowledge of drug levels or status of anti-drug antibodies
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Therapeutic drug monitoring — Treatment algorithm based on assessments of serum drug levels and anti-drug antibodies
  Arms: Therapeutic drug monitoring
Other: Standard care — Treatment algorithm based on standard clinical assessments, without knowledge of serum drug levels and anti-drug antibodies
  Arms: Standard care

SUMMARY:
Infliximab and other TNF-inhibitors have revolutionised the treatment of several immunological inflammatory diseases. Still, more than half of the patients either do not respond sufficiently to infliximab therapy or loose efficacy over time. The large individual variation in the serum drug concentrations on standard doses and the development of anti-drug antibodies are thought to be main reasons for these treatment failures. An individualised treatment strategy based on systematic assessments of serum drug concentrations, therapeutic drug monitoring, has been proposed as a clinical tool to optimise efficacy of infliximab treatment. Therapeutic drug monitoring seems reasonable both from a clinical and an economical point of view, but the effectiveness of this treatment strategy still remain to be shown. The NOR-DRUM study is planned as a national, randomised controlled multicentre trial in two parts aiming to assess the effectiveness of therapeutic drug monitoring in order to achieve remission in patients with immunological inflammatory diseases starting infliximab treatment (part A) and in order to maintain disease control in patients on maintenance infliximab treatment (part B). The results of the NOR-DRUM study will hopefully contribute to an implementation of a personalised medicine approach to treatment with infliximab and other biological drugs.

ELIGIBILITY:
Inclusion Criteria:

NOR-DRUM A

1. A clinical diagnosis of one of the following; rheumatoid arthritis, spondyloarthritis (including ankylosing spondylitis), psoriatic arthritis*, ulcerative colitis, Crohn's disease or chronic plaque psoriasis
2. Male or non-pregnant female
3. ≥18 and < 75 years of age at screening
4. A clinical indication to start INX
5. Subject not in remission according to diagnosis-specific disease activity scores
6. Subject capable of understanding and signing an informed consent form

   * Patients with psoriatic arthritis with predominantly axial manifestations should be included and assessed as spondyloarthritis

NOR-DRUM B

1. A clinical diagnosis of one of the following; rheumatoid arthritis, spondyloarthritis (including ankylosing spondylitis), psoriatic arthritis*, ulcerative colitis, Crohn's disease or chronic plaque psoriasis
2. Male or non-pregnant female
3. ≥18 and < 75 years of age at screening
4. On maintenance therapy with infliximab for a minimum of 30 weeks and a maximum of 3 years
5. A clinical indication for further infliximab treatment
6. Subject capable of understanding and signing an informed consent form

   * Patients with psoriatic arthritis and predominantly axial manifestations should be included and assessed as spondyloarthritis

Exclusion Criteria:

NOR-DRUM A

1. Major co-morbidities, such as previous malignancies within the last 5 years, severe diabetes mellitus, severe infections (including HIV), uncontrollable hypertension, severe cardiovascular disease (NYHA class 3 or 4), severe respiratory diseases, demyelinating disease, significant chronic widespread pain syndrome, laboratory abnormalities or significant renal or hepatic disease and/or other diseases or conditions where treatment with infliximab is either found contra-indicated by the clinician or which make adherence to the protocol difficult
2. A positive screening for TB and hepatitis
3. Inadequate birth control, pregnancy or subject considering becoming pregnant during the study period
4. Psychiatric or mental disorders, alcohol abuse or other substance abuse, language barriers or other factors which makes adherence to the study protocol difficult
5. Prior use of infliximab within the last 6 months

NOR-DRUM B

1. Major co-morbidities, such as previous malignancies within the last 5 years, severe diabetes mellitus, severe infections, uncontrollable hypertension, severe cardiovascular disease (NYHA class 3 or 4), severe respiratory diseases, demyelinating disease, significant chronic widespread pain syndrome, laboratory abnormalities or significant renal or hepatic disease and/or other diseases or conditions where treatment with infliximab is either found contra-indicated by the clinician or which make adherence to the protocol difficult
2. Inadequate birth control, pregnancy or subject considering becoming pregnant during the study period
3. Psychiatric or mental disorders, alcohol abuse or other substance abuse, language barriers or other factors which makes adherence to the study protocol difficult

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 611 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2020-12-14 (Actual)

PRIMARY OUTCOMES:
Proportion of patients in remission defined by disease specific composite scores Study part A | 30 weeks
  Definition of remission: DAS 28 score <2.6 in patients with RA and PsA, ASDAS score <1.3 in patients with SpA, Mayo score of ≤2 with no sub scores >1 in patients with UC, HBI score of ≤4 in CD and PASI score of ≤4 in patients with Ps.
Sustained disease control throughout the study period without disease worsening defined by disease specific composite scores Study part B | 52 weeks
  Definition of disease worsening: RA/PsA: Change DAS28 of ≥ 1.2 and min DAS 3.2 SpA: Increase in ASDAS of ≥1.1 and min ASDAS of 2.1 UC: Increase in Partial Mayo score of ≥ 3 and min score of ≥ 5 CD: Increase in HBI of ≥ 4 points and min score of 7 Ps: Increase in PASI of ≥ 3 points and min PASI score of 5 Or: Patient and investigator consensus on disease worsening

SECONDARY OUTCOMES:
Time to sustained remission (Part A) | Assessed at all time points up to 30 weeks
  Remission at all following visit
Patient's and physician's global assessment of disease activity (Part A and B) | 30 weeks (A) and 52 weeks (B)
  Visual analogue scale (VAS) 0 mm-100 mm (100 mm worst outcome)
ESR (Part A and B) | 30 weeks (A) and 52 weeks (B)
  0-100 mmHg
CRP (Part A and B) | 30 weeks (A) and 52 weeks (B)
  mg/L
Occurrence of anti-drug antibodies (Part A and B) | 30 weeks (A) and 52 weeks (B)
  Defined as ADAb ≥15 µg/L
Occurrence of drug discontinuation (Part A and B) | 30 weeks (A) and 52 weeks (B)
  Infliximab discontinuation
Cost effectiveness, QALY | 30 weeks (A) and 52 weeks (B)
  Part A and B (Incremental Quality adjusted life years (QALYs) of the intervention arm and active comparator)
Cost effectiveness, ICERs | 30 weeks (A) and 52 weeks (B)
  Part A and B (Cost-effectiveness ratios (ICERs) of the intervention arm and active comparator)
Health utility (EQ-5D) | 30 weeks (A) and 52 weeks (B)
  EuroQol 5 (EQ-5D) dimensions The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state
Quality of life (SF-36) | 30 weeks (A) and 52 weeks (B)
  The SF-36 is a multi-purpose, short-form health survey with 36 questions. The SF-36 will be scored according to RAND 36-Item Health Survey 1.0 to form eight measures scores 0-100 (100 worst outcome): physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions.
Safety (adverse events frequency) | 30 weeks (A) and 52 weeks (B)
  A and B
Time to disease worsening | 52 weeks
  Part B
Proportion of patients in remission, diagnostic subgroups (overall in B) | 30 weeks (A) and 52 weeks (B)
  RA/PsA: DAS28 remission, SDAI remission, ACR/EULAR remission, SpA: ASDAS inactive disease, UC: PMS, CD: HBI, Ps PASI
Serum drug level | Assessed at all time points up to 30 weeks
  Trough level
Proportion of patients with improvement defined by disease specific composite scores (Part A) | 14 weeks
  * Improvement in RA and PsA Improvement is defined as a decrease in DAS28 of ≥1.2 from baseline
  * Improvement in SpA Improvement is defined as a decrease in ASDAS of ≥1.1 from baseline
  * Improvement in UC Improvement in UC is defined as a decrease in the partial Mayo score of ≥ 3 points from baseline or a partial Mayo score of 0
  * Improvement in CD Improvement in CD is defined as a decrease in HBI of ≥ 4 points from baseline
  * Improvement in Ps Improvement in Ps is defined as PASI 50 (A 50% decrease in the PASI obtained at baseline)
  * Patient and investigators consensus on improvement
Time to remission (Part A) | Assessed at all time points up to week 30
  Definition of remission: DAS 28 score <2.6 in patients with RA and PsA, ASDAS score <1.3 in patients with SpA, Mayo score of ≤2 with no sub scores >1 in patients with UC, HBI score of ≤4 in CD and PASI score of ≤4 in patients with Ps.
DAS28 (RA and PsA only) | 30 weeks (A) and 52 weeks (B)
  The 28-joint Disease Activity Score (DAS28) includes the 28- tender joint counts (TJC28), 28-swollen joint counts (SJC28), Erythrocyte Sedimentation Rate (ESR) and Patient Global Assessment (PGA) on a VAS
  According to DAS28, the following cut-points are used:
  High disease activity: DAS28 > 5.1 Moderate disease activity: 5.1 ≥ DAS28>3.2 Low disease activity: 3.2 ≥ DAS28 ≥ 2.6 In remission: DAS28 < 2.6
Partial Mayo score | 30 weeks (A) and 52 weeks (B)
  The Mayo score consists of four components (rectal bleeding, stool frequency, physician rating of disease activity, and mucosal appearance at endoscopy) rated from 0-3 that are summed to give a total score that ranges from 0-12. The non-invasive partial Mayo score (PMS) does not require an endoscopy, and thereby ranging from 0-9.
  Remission is defined as a partial Mayo score of ≤ 2 with no individual subscore >1
SDAI (RA and PsA only) | 30 weeks (A) and 52 weeks (B)
  The Simplified Disease Activity Index (SDAI) includes TCJ28, SJC28, PGA, PhGA and CRP. In remission: SDAI ≤ 3.3. High values denotes worse outcomes. High values denotes worse outcomes.
EULAR response (RA and PsA only) | 30 weeks (A)
  Defined according to EULAR definition
ACR/EULAR remission | 30 weeks (A)
  * TJC28 ≤ 1
  * SJC28 ≤ 1
  * CRP ≤ 10 (mg/l)
  * PGA ≤ 14
ACR response | 30 weeks (A)
  If a patient experiences a flare and treatment is escalated, the ACR response rates ACR20, ACR50, ACR70 and ACR90 as well as ACR remission rates will be calculated.
  An ACR20 response is defined if the following criteria are fulfilled:
  * 20% improvement in RAI AND
  * 20% improvement in swollen joint count 44 AND
  * 20% improvement in at least 3 of 5 other core set items
  The other core set items consist of:
  * Investigator global assessment of disease activity
  * Patient global assessment of disease activity
  * Patient pain
  * Disability
  * ESR/CRP
DAPSA (PsA only) | 30 weeks (A) and 52 weeks (B)
  Disease Activity index for PSoriatic Arthritis (DAPSA) is calculated as follows: TJC68 + SJC66 + CRP(mg/L)/10 + PGA(0-100)/10+VAS Pain(0-100)/10. High values denotes worse outcomes.
BASDAI (SpA only) | 30 weeks (A) and 52 weeks (B)
  The Bath Ankylosing Spondylitits Disease Activity Index (BASDAI) includes six questions pertaining to the five major symptoms of ankylosing spondylitis: fatigue (Q1), spinal pain (Q2), joint pain/swelling (Q3), areas of localized tenderness (Q4), morning stiffness duration (Q5) and morning stiffness severity (Q6). Each question is scored on an NRS (0-10).
ASDAS | 30 weeks (A) and 52 weeks (B)
  The Ankylosing Spondylitis Disease Activity Score (ASDAS) is computed based on patient reported outcomes (components of BASDAI) and the CRP. The ASDAS-CRP is calculated as follows:
  ASDAS-CRP=0.121*total back pain + 0.0110*patient global + 0.073*peripheral pain/swelling + 0.058*duration of morning stiffness + 0.579*ln(CRP+1 High values denotes worse outcomes
Partial Mayo Score (UC only) | 30 weeks (A) and 52 weeks (B)
  The Mayo score consists of four components (rectal bleeding, stool frequency, physician rating of disease activity, and mucosal appearance at endoscopy) rated from 0-3 that are summed to give a total score that ranges from 0-12. The non-invasive partial Mayo score (PMS) does not require an endoscopy, and thereby ranging from 0-9.
  Remission is defined as a partial Mayo score of ≤ 2 with no individual subscore >1
Harvey-Bradshaw Index (CD only) | 30 weeks (A) and 52 weeks (B)
  The Harvey-Bradshaw index (HBI) consists of five domains, general well-being (0-4), abdominal pain (0-3), number of liquid soft stools per day, abdominal mass (0-3) and number of predefined complications. The scores of each sub-domain is summed up to compute the HBI.
  Remission is defined as a HBI score ≤ 4 points.
Psoriasis Area and Severity Index (PASI) (Ps only) | 30 weeks (A) and 52 weeks (B)
  A PASI 50/75 means a 50% /75% reduction in the PASI score. Complete clearance is defined as PASI=0, mild to moderate psoriasis is defined as PASI < 10, moderate to severe psoriasis between 10 and 20 and severe psoriasis above 20.
  Remission is defined as PASI <4
Modified Health Assessment Questionnaire | 30 weeks (A) and 52 weeks (B)
  Each item of the Modified Health Assessment Questionnaire (MHAQ) is scored on a categorical 0-3 scale and the sum score is divided by 8 to form the MHAQ score 0.0 to 3.0 (3.0 worst outcome possible)
Rheumatoid Arthritis Impact of Disease (RA only) | 30 weeks (A) and 52 weeks (B)
  The Rheumatoid Arthritis Impact of Disease (RAID) score is calculated based on seven numerical rating scales (NRS) questions. Each NRS is assessed as a number between 0 and 10. The seven NRS correspond to pain, function, fatigue, sleep, emotional wellbeing, physical wellbeing and coping/self-efficacy.
Psoriatic Arthritis Impact of Disease (PsAID) score | 30 weeks (A) and 52 weeks (B)
  Psoriatic Arthritis Impact of Disease (PsAID) score is a questionnaire with 9 domains of health. The nine domains with relative weights are: pain (0.174), fatigue (0.131), skin (0.121), work and/or leisure activities (0.110), function (0.107), discomfort (0.098), sleep (0.089), coping (0.087) and anxiety (0.085), each rated on an NRS (0-10). The rates of each domain are weighted and summed to form a score in the range of 0-10 (10 worst outcome possible). The final RAID score is computed. The scale 0-10 where higher figures indicate worse status.
Inflammatory Bowel Disease Questionnaire (IBDQ) | 30 weeks (A) and 52 weeks (B)
  The Inflammatory Bowel Disease Questionnaire (IBDQ) is widely used tool to measure health-related quality of life in patients with inflammatory bowel diseases. The questionnaire consists of 32 questions scored in four domains: bowel symptoms, emotional health, systemic systems and social function. The total IBDQ score is the sum of all the question scores, ranging 32 to 224 (224 worst possible)
Total drug consumption | 30 weeks (A) and 52 weeks (B)
  mg/kg/ week
Dermatology Life Quality Index (DLQI) | 30 weeks (A) and 52 weeks (B)
  The Dermatology Life Quality Index (DLQI) consists of 10 questions concerning patients' perception of the impact of skin diseases on different aspects of their health-related quality of life over the last week. It has been validated for adult dermatology patients aged 16 years and older. The items of the DLQI encompass aspects of symptoms and feelings, daily activities, leisure, work or school, personal relationships and the side effects of treatment. Each question is scored on a 4-point Likert scale: Not at all/Not relevant=0, A little=1, A lot=2 and Very much=3. Scores of individual items (0-3) are added to yield a total score (0-30); higher scores mean greater impairment of patient's QoL. The DLQI will only be presented to patients with chronic plaque psoriasis.
Calprotectin | 30 weeks (A) and 52 weeks (B)
  Faecal calprotectin is an inflammatory marker for IBD. It is measured in mg/kg

CONTACTS AND LOCATIONS:
Overall Officials: Espen A Haavardsholm, MD, PhD, Principal Investigator — Diakonhjemmet Hospital; Tore K Kvien, MD, PhD, Study Director — Diakonhjemmet Hospital
Locations (21):
- Norway (21):
  - Akershus University Hospital, Oslo, Lørenskog
  - Sørlandet Sykehus, Arendal, Arendal
  - Ålesund, HELSE MØRE OG ROMSDAL HF, Ålesund
  - Haukeland, HELSE BERGEN HF,, Bergen
  - Bodø, NORDLANDSSYKEHUSET, Bodø
  - Drammen, VESTRE VIKEN HF, Drammen
  - Elverum, SYKEHUSET INNLANDET HF, Elverum
  - Helse Førde Hf, Førde
  - Hamar, SYKEHUSET INNLANDET HF, Hamar
  - HAUGESUND SANITETSFORENING revmatismesykehus, Haugesund
  - Haugesund Sjukehus, Haugesund
  - SØRLANDET SYKEHUS HF Kristiansand, Kristiansand
  - REVMATISMESYKEHUSET AS, Lillehammer, Lillehammer
  - Sykehuset Østfold Moss, Moss
  - Rikshospitalet, Oslo
  - Diakonhjemmet Sykehus, Oslo
  - Betanien Hospital, Skien
  - Stavanger Universitetssjukehus, Stavanger
  - Tromsø, UNIVERSITETSSYKEHUSET NORD-NORGE HF, Tromsø
  - St Olavs Hospital, Trondheim
  - Sykehuset Vestfold, Tønsberg, Tønsberg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Syversen SW, Jorgensen KK, Goll GL, Brun MK, Sandanger O, Bjorlykke KH, Sexton J, Olsen IC, Gehin JE, Warren DJ, Klaasen RA, Noraberg G, Bruun TJ, Dotterud CK, Ljosa MKA, Haugen AJ, Njalla RJ, Zettel C, Ystrom CM, Bragnes YH, Skorpe S, Thune T, Seeberg KA, Michelsen B, Blomgren IM, Strand EK, Mielnik P, Torp R, Mork C, Kvien TK, Jahnsen J, Bolstad N, Haavardsholm EA. Effect of Therapeutic Drug Monitoring vs Standard Therapy During Maintenance Infliximab Therapy on Disease Control in Patients With Immune-Mediated Inflammatory Diseases: A Randomized Clinical Trial. JAMA. 2021 Dec 21;326(23):2375-2384. doi: 10.1001/jama.2021.21316. PMID 34932077
- [Derived] Syversen SW, Goll GL, Jorgensen KK, Sandanger O, Sexton J, Olsen IC, Gehin JE, Warren DJ, Brun MK, Klaasen RA, Karlsen LN, Noraberg G, Zettel C, Ljosa MKA, Haugen AJ, Njalla RJ, Bruun TJ, Seeberg KA, Michelsen B, Strand EK, Skorpe S, Blomgren IM, Bragnes YH, Dotterud CK, Thune T, Ystrom CM, Torp R, Mielnik P, Mork C, Kvien TK, Jahnsen J, Bolstad N, Haavardsholm EA. Effect of Therapeutic Drug Monitoring vs Standard Therapy During Infliximab Induction on Disease Remission in Patients With Chronic Immune-Mediated Inflammatory Diseases: A Randomized Clinical Trial. JAMA. 2021 May 4;325(17):1744-1754. doi: 10.1001/jama.2021.4172. PMID 33944876
- [Derived] Syversen SW, Goll GL, Jorgensen KK, Olsen IC, Sandanger O, Gehin JE, Warren DJ, Sexton J, Mork C, Jahnsen J, Kvien TK, Bolstad N, Haavardsholm EA. Therapeutic drug monitoring of infliximab compared to standard clinical treatment with infliximab: study protocol for a randomised, controlled, open, parallel-group, phase IV study (the NOR-DRUM study). Trials. 2020 Jan 6;21(1):13. doi: 10.1186/s13063-019-3734-4. PMID 31907007